CLINICAL TRIAL: NCT00780026
Title: Effect Of Intraoperative Strict Glycemic Control During Liver Transplantation On Postoperative Morbidity And Mortality
Brief Title: Intraoperative Glucose Control in Liver Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shawn J. Pelletier, MD, Associate Professor of Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00016106
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Liver Transplant
Keywords: liver; transplant; blood sugar
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Strict Glycemic Control (Experimental): strict glycemic control (80 to 110 mg/dl)
  Interventions: Drug: insulin
- Standard of Care Control (No Intervention): standard of care insulin dosing

INTERVENTIONS:
Drug: insulin — bolus or infusion 80 to 110 mg/dl
  Arms: Strict Glycemic Control

SUMMARY:
The goal of the proposed study is to evaluate the effectiveness of intraoperative, strict glycemic control to improve survival and infection rates following liver transplantation in a randomized, prospective trial.Primary objective: To determine if strict intraoperative blood glucose control, when compared to standard intraoperative glycemic control, improves 1-year recipient survival and decreases surgical complications, including infections, following liver transplantation.

DETAILED DESCRIPTION:
Approximately 2.1 million patients in the United States acquire infections during medical care every year. For example, 9%-30% patients who undergo surgery acquire nosocomial infections, which increase mortality and morbidity over that expected normally expected and increase the cost of care by several billion dollars. Studies have shown that controlling high blood glucose levels dramatically improves the recovery of critically ill patients after surgery, most notably decreasing the risk of infection. The advantage of strict glycemic control in the critically ill patient is now well accepted, and the Institute for Healthcare Improvement and Surviving Sepsis Campaign set glycemic control as part of the post-operative sepsis management bundle.

Few studies have investigated the role of strict glycemic control during surgery itself. Liver transplantation is a good model for studying glucose control as hyperglycemia almost always occurs and the incidence of infection is higher than with other surgical procedures. We performed a retrospective review of 184 consecutive adult liver recipients in which intra-operative blood glucose levels were measured and treated with insulin. Recipients with strict glycemic control were compared to those with poor control for differences in donor and recipient demographics, intra-operative blood glucose concentrations, intra-operative insulin administered, immunosuppression, post-operative complications, and mortality. Poor glycemic control was associated with a significantly increased rate of infection during the first 30 days post-operatively (48% vs. 33%, P=0.05) and 1-year mortality was significantly increased for those recipients with poor intra-operative glucose control (21.9% vs. 8.8%; P = 0.05). These data along with the post-operative studies, suggest that the post-transplant mortality rate may potentially be decreased by nearly 50% at 1 year and underscore the need for this to be confirmed in a prospective trial.

The goal of this study is to prospectively evaluate the outcomes of liver transplant recipients to either strict glucose control (goal of 80-110 mg/dl) or the current standard of care (goal of between 180 and 200 mg/dl). The specific aim of this study is to determine if strict intra-operative blood glucose control, improves 1-year recipient survival and decreases surgical complications, including infections, following liver transplantation. The rates of infection at 30 days after surgery and health at one year post- surgery will be compared. The frequency of other common post-operation complications will also be studied. The proposed study has the potential to have an impact on the intra-operative management of all liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years old undergoing liver transplantation
* Patients willing and capable of giving written informed consent for study participation

Exclusion Criteria:

* Multi-organ transplant recipients
* Patients receiving a liver incompatible with A, B or O blood types
* HIV infected patients
* Recipients of an organ from an HIV+ donor
* Patients with severe coexisting disease or presenting with any unstable medical condition which could affect the study objectives
* Patients with a co-existing alcoholic disease who have not been abstinent for at least 6 month immediately prior to transplantation and are not expected to be able to remain abstinent after transplantation
* Patients who are unlikely to comply with the study requirements or unable to give informed consent
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer or if such therapy is to be instituted posttransplantation
* Patients transplanted for hepatocellular carcinoma exceeding 3 nodules or with nodule diameter larger than 5 cm
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadatropin (hCG) laboratory test (> 5 milli-International units (mIU/ml)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Pelletier, MD, Principal Investigator — Universitry of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Kumar SS, Pelletier SJ, Shanks A, Thompson A, Sonnenday CJ, Picton P. Intraoperative glycemic control in patients undergoing Orthotopic liver transplant: a single center prospective randomized study. BMC Anesthesiol. 2020 Jan 4;20(1):3. doi: 10.1186/s12871-019-0918-0. PMID 31901245

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Strict Glycemic Control | Standard of Care Control
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strict Glycemic Control | Standard of Care Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [48 to 57] | 55 [50.0 to 59.0] | 54 [49.0 to 59.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 36 | 74
  Male | 12 | 14 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 41 | 41 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 41 | 41 | 82
  African American | 5 | 4 | 9
  Asian | 0 | 1 | 1
  Other | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100
BMI [Median (Inter-Quartile Range); unit: kg/m2] — The BMI is defined as the body mass (in kilograms) divided by the square of the body height (in meters).
  kg/m2 | 30.4 [25.7 to 35.9] | 28.9 [25 to 32.4] | 29.6 [25.1 to 34.0]
Pre-existing conditions [Count of Participants; unit: Participants] — Preexisting diagnosis for Coronary Artery Disease (CAD)
  Participants
    Diabetes | 13 | 16 | 29
    Coronary Artery Disease(CAD) | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Infection Rates
Description: Number of participants who sustained an infection after surgery
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Strict Glycemic Control | Standard of Care Control
Number analyzed (Participants) | 50 | 50
Participants
  Bacterial Infection | 27 | 26
  Fungal Infection | 11 | 7
  Transplant Incision wound | 9 | 7
  Viral | 4 | 6
Statistical Analysis 1: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.841, Chi-squared — P value for Bacterial infection
Statistical Analysis 2: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.298, Chi-squared — P-value for fungal infection
Statistical Analysis 3: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.585, Chi-squared — P value for transplant incision wound
Statistical Analysis 4: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.505, Chi-squared — P value for viral infection

2. Primary Outcome: Number of Participants With One Year Survival Post Transplant
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Strict Glycemic Control | Standard of Care Control
Number analyzed (Participants) | 50 | 50
Participants | 44 | 44
Statistical Analysis 1: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.999, Fisher Exact

3. Secondary Outcome: Hospital Length of Stay
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Strict Glycemic Control | Standard of Care Control
Number analyzed (Participants) | 50 | 50
days | 12.5 [8 to 19] | 11 [8 to 19]
Statistical Analysis 1: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Equivalence — If the p-value for the means is > 0.05 between the groups then they will be deemed equivalent; p = 0.384, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Participants Who Required Postoperative Blood Transfusion Within 3 Days in the ICU
Description: Requirements for blood transfusion counted as a binary variable yes/no per participant
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Strict Glycemic Control | Standard of Care Control
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With a Need for Hemodialysis
Description: Number of people who had renal failure in the year following liver transplant and needing hemodialysis to support it;
Time Frame: 12 months post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Strict Glycemic Control | Standard of Care Control
Number analyzed (Participants) | 50 | 50
Participants | 6 | 9
Statistical Analysis 1: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.401, Fisher Exact

6. Secondary Outcome: Number of Participants With Biliary Complications
Description: Number of participants who experienced bile leak or biliary Stricture
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Strict Glycemic Control | Standard of Care Control
Number analyzed (Participants) | 50 | 50
Participants
  bile leak | 14 | 15
  Biliary Stricture | 13 | 20
Statistical Analysis 1: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.826, Chi-squared — P value for bile leak
Statistical Analysis 2: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.137, Chi-squared — This is the p value for Biliary Stricture

7. Secondary Outcome: Number of Participants With Venous Thrombotic Complications
Description: Number of participants who were diagnosed with portal vein thrombosis post surgery
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Strict Glycemic Control | Standard of Care Control
Number analyzed (Participants) | 50 | 50
Participants | 3 | 3
Statistical Analysis 1: Comparison: Strict Glycemic Control vs Standard of Care Control; Test type: Superiority or Other; p = 0.999, Fisher Exact

ADVERSE EVENTS:
Time Frame: All cause mortality and graft loss were followed for 5 years, whereas all other adverse events were followed for 30 days.
Arm/Group | Strict Glycemic Control | Standard of Care Control
All-Cause Mortality (participants affected / at risk) | 12/50 | 9/50
Serious Adverse Events (participants affected / at risk) | 16/50 | 11/50
Other Adverse Events (participants affected / at risk) | 45/50 | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Strict Glycemic Control (N=50) | Standard of Care Control (N=50)
Graft Loss (Hepatobiliary disorders) | 16 | 11 — Liver
Death (Hepatobiliary disorders) | 12 | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Strict Glycemic Control (N=50) | Standard of Care Control (N=50)
Infections (Infections and infestations) | 35 | 32 — Combination of bacterial, fungal, transplant incision wound or viral infections
Bile Leak (Hepatobiliary disorders) | 14 | 15
Biliary Stricture (Hepatobiliary disorders) | 13 | 20
Major Cardiac Event (Cardiac disorders) | 4 | 5
Portal Vein Thrombosis (Vascular disorders) | 3 | 3
Re-operation for bleeding (Surgical and medical procedures) | 10 | 6
Re-operation - other (Surgical and medical procedures) | 15 | 9
Dialysis - renal failure (Renal and urinary disorders) | 6 | 9
Wound dehiscence (Surgical and medical procedures) | 12 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes